CLINICAL TRIAL: NCT00989430
Title: Prism Adaptation Therapy for Spatial Neglect: Theoretical and Practical Outcomes
Brief Title: Prism Adaptation Therapy for Spatial Neglect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, A. M. Barrett, MD, Director, Stroke Rehabilitation Research, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMBarrett3; Spatial Neglect (Other Grant/Funding Number: NIDRR H133G120203)
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Spatial Neglect; Deficits in Attention Motor Control and Perception
Keywords: stroke; CVA; cerebrovascular accident; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prism Adaptation Treatment (Experimental): Two weeks of prism adaptation treatment followed by 4 weekly assessments and long-term follow-ups at the 3rd and 6th months.
  Interventions: Behavioral: Prism Adaptation Treatment
- Control: Standard Rehabilitation Care (No Intervention): Participants will continue with their standard inpatient rehabilitation care. They will be assessed with cognitive and functional scales for tracking their recovery.

INTERVENTIONS:
Behavioral: Prism Adaptation Treatment — Wearing prism goggles and performing visuomotor tasks during therapy sessions.
  Arms: Prism Adaptation Treatment

SUMMARY:
The purpose of this research study with a randomized controlled design is to examine the effects of prism adaptation treatment on two visual-spatial recovery components. After a stroke, an "internal GPS", locating where objects or people lie in a particular area of space, may be impaired. Alternately, a stroke may impair precise visual-spatial hand and body aiming movements. The research team wishes to discover whether prism adaptation treatment (two weeks of daily 20-min sessions of goal-directed movement with prism goggles) affects visual-spatial where or aiming errors selectively after stroke.

This research represents one of the first attempts to apply what we know about the brain from neuroscience research, to modern clinical rehabilitation practices.

DETAILED DESCRIPTION:
The purpose of this research study with a randomized controlled design is to examine the effects of prism adaptation treatment on two visual-spatial recovery components. After a stroke, an "internal GPS", locating where objects or people lie in a particular area of space, may be impaired. Alternately, a stroke may impair precise visual-spatial hand and body aiming movements. The research team wishes to discover whether prism adaptation treatment (two weeks of daily 20-min sessions of goal-directed movement with prism goggles) affects visual-spatial where or aiming errors selectively after stroke.

This research represents one of the first attempts to apply what we know about the brain from neuroscience research, to modern clinical rehabilitation practices.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 to 100 years of age, inclusive.
* The subject has had a stroke on the right side of the brain.
* The subject is able to give Informed consent.
* The subject has a spatial neglect (if known).
* The subject is able and willing to comply with the study protocol, including availability for all scheduled clinic visits.

Exclusion Criteria:

* The subject has or had a serious brain condition other than stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-10; Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Kessler Foundation Neglect Assessment Process | 6 months
  a performance based and behavioral measure for spatial neglect that utilizes and standardizes the administration of the Catherine Bergego Scale (CBS)

SECONDARY OUTCOMES:
Behavior Inattention Test | 2 weeks
  Conventional subtest, a set of paper and pencil test for spatial neglect
Barthel Index | 2 weeks
  A functional independence assessment of daily tasks

CONTACTS AND LOCATIONS:
Overall Officials: A. M. Barrett, MD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States

REFERENCES:
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963
- [Derived] Boukrina O, Chen P, Budinoska T, Barrett AM. Exploratory examination of lexical and neuroanatomic correlates of neglect dyslexia. Neuropsychology. 2020 May;34(4):404-419. doi: 10.1037/neu0000619. Epub 2020 Jan 30. PMID 31999167
- [Derived] Caulfield MD, Chen P, Barry MM, Barrett AM. Which perseverative behaviors are symptoms of spatial neglect? Brain Cogn. 2017 Apr;113:93-101. doi: 10.1016/j.bandc.2016.11.002. Epub 2017 Feb 3. PMID 28167411
- See also: Kessler Foundation Stroke Program — https://kesslerfoundation.org/researchcenter/stroke/index.php